CLINICAL TRIAL: NCT05645588
Title: Pranayama for Outpatients With Posttraumatic Stress Disorder: a Randomized-controlled Trial
Brief Title: Pranayama for Posttraumatic Stress Disorder
Acronym: PRANAPTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no sufficient funding, employee have left the company
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Director of Research, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-10859-BO
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Pranayama; Yoga; Complimentary Therapies; Somatic Symptom Disorder; SSD; PTSD; Safety; Effectiveness; Randomized Controlled Trail
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and Therapists (Care Provider) could not be blinded according to the nature of the intervention. However, therapists will be blinded to allocation concealment as they do not be aware of the patients' group assignment at baseline assessment until they open the opaque randomization envelope, which contains the patient randomization number and group assignment. The random sequence generation and the envelopes were prepared by the study coordinator who is not involved patient recruitment. Patients received post intervention questionnaires from a study assistant/nurse of the respective outpatient department (outcome assessor) who is also blinded to the patients' group assignment. After completing the questionnaires, the study assistant will sent them to study coordinator so that the therapist could not influence the patients' answers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pranayama assisted trauma-focused standard psychotherapy (TF-SPT). (Experimental): Behavioral: Pranayama assisted trauma-focused standard psychotherapy (TF-SPT) The pranayama intervention is placed directly at the begin of the respective TF-SPT unit and will be repeated for 10 subsequent TF-SPT units.
  Interventions: Behavioral: Pranayama assisted trauma-focused standard psychotherapy (TF-SPT)
- Trauma-focused standard psychotherapy (TF-SPT) (Active Comparator): Behavioral: Patients wait for 10 TF-SPT units and then are offered to learn pranayama.
  Interventions: Behavioral: Trauma-focused standard psychotherapy (TF-SPT)

INTERVENTIONS:
Behavioral: Pranayama assisted trauma-focused standard psychotherapy (TF-SPT) — To prepare patients for the TF-SPT, they received 5-10 minutes of pranayama at the begin of each of the 10 TF-SPT units.
  Arms: Pranayama assisted trauma-focused standard psychotherapy (TF-SPT).
Behavioral: Trauma-focused standard psychotherapy (TF-SPT) — Patients wait for 10 TF-SPT units and then are offered to learn pranayama
  Arms: Trauma-focused standard psychotherapy (TF-SPT)

SUMMARY:
This study aims to investigate the effect of pranayama (yoga-breathing techniques) on post-traumatic symptom severity in patients with post-traumatic stress disorder undergoing standard, out-patient, trauma-focused psychotherapy. Therefore, short pranayama sessions of 5-10 minutes will be provided to the patients directly at the begin of each of psychotherapy unit, while the control group will receive standard, trauma-focused psychotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PTSD according to ICD-10 F43.1
* PCL-5 Score of at least 33 points
* Undergoing outpatient standard trauma-focused psychotherapy (Cognitive Behavioral Therapy, Psychodynamic Psychotherapy, or Systemic Psychotherapy)

Exclusion Criteria:

* Pre-existing mental or somatic conditions that are unlikely to result in correct or safe performance of pranayama:

  1. Substance dependence current use (ICD-10 F10.X, F11.X).
  2. Dementia (ICD-10 F00-F03)
  3. Somatoform Disorder (ICD F45.X) of moderate or severe degree according to DSM-5 300.82: ≥ 2 reactions (cognitive, emotional, or behavioral) to somatic symptoms (≥ 2 criterion-B)
  4. Severe cardiovascular disease: presence of cardiac or vascular implants or grafts, e.g., pacemaker (ICD-10 Z95.X), condition after organ or tissue transplantation (ICD-10 Z94.X)
  5. Acute adverse events occurring during pranayama at baseline (including neck pain, subjective sensation of pressure in the lungs, anxiety / panic)
* Cancer diagnosis in the past 5 years (ICD-10 C00-C97, D37-48)
* Pregnancy / breastfeeding
* Regular pranayama practice in the last 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of posttraumtic symptoms | week 10
  Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): The PCL-5 is a standard 20-item scale with a sum score ranging from 0 to 80 points. The cut-off point for clinically relevant symptom severity is 33 points.

SECONDARY OUTCOMES:
Health-related quality of life | week 10
  Short Form 12 Health Survey (SF-12): The SF-12 is a standard 12-item scale with two sum scores (physical and mental quality of life) ranging from 0 to 100 points.
Anxiety | week 10
  Beck Anxiety Inventory (BAI): The BAI is a standard 21-items scale ranging from 0 to 63 points with 0-7 points = minimal anxiety, 8-15 points = mild anxiety, 16-25 points = moderate anxiety, and 26-63 points = clinically relevant anxiety.
Depression | week 10
  Beck Depression Inventory Revision (BDI-II): The BDI-II is a standard 21-items scale ranging from 0 to 63 points with 0-13 points =no/clinically not relevant depression/depression in remission, 14-19 points = mild depression, 20-28 points = moderate depression und 29-63 points = severe depression.
Breath Holding Duration | week 10
  Breath Holding Task (BHT): The BHT is standard test procedure for the measurement of ability of the suppression of the respiratory reflex.
Adverse Events | weeks 1,2,3,4,5,6,7,8,9,10
  Number of patients with adverse events and types of the adverse events
Therapist Global Improvement | week 10
  Clinician Global Impression of Improvement (CGI-I) rated by the therapist on 1 item ranging from 1 to 7.
Patient Global Improvement | week 10
  Patient Global Impression of Improvement (PGI-I) rated by the patient on 1 item ranging from 1 to 7.

OTHER OUTCOMES:
Treatment Expectation | week 0
  Treatment Credibility Scale (TCS): The TCS is a standard NRS scale ranging from 0 points (lowest expectation of treatment effectiveness) to 10 points (highest expectation of treatment effectiveness).
Interoceptive Awareness | weeks 0+10
  Multidimensional Assessment of Interoceptive Awareness, Version 2 (MAIA-II): The MAIA-II is a 37-item questionnaire. It includes 8 subscales. Scores ranged between 0 and 5, where higher score indicate more awareness of bodily sensation. Percentiles can also be calculated, indicating how the score is associated to a normative sample.
Social Readjustment after life events | weeks 0+10
  Social Readjustment Rating Scale (SRRS): The SRRS consists of 43 items. A sum score of 1-149 = low stress level; 150-299 = 30% probability of developing a stress-associated disease; 300 and more = 80% probability of developing a stress-associated disease.
Compliance | weeks 0,1,2,3,4,5,6,7,8,9,10
  Diary (via App): daily pranayama practice, BHT time
Medication | weeks 0+10
  A change in medication between weeks 0 and 10 is recorded.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code